CLINICAL TRIAL: NCT00524485
Title: A Pilot Study to Investigate the Use of Topical Levulan® With Vbeam® Laser for the Treatment of Actinic Keratoses
Brief Title: Photodynamic Therapy Using Topical Aminolevulinic Acid in Treating Patients With Actinic Keratosis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Withdrawn due to low accrual
Sponsor: Roswell Park Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I 28204; RPCI-I-28204
Record Dates: First submitted 2007-08-31; First posted 2007-09-03 (Estimated); Results first posted 2017-05-17 (Actual); Last update posted 2017-06-14 (Actual); Status verified 2017-05

CONDITIONS: Precancerous/Nonmalignant Condition
Keywords: actinic keratosis
MeSH Terms: conditions — Precancerous Conditions; Keratosis, Actinic | interventions — Aminolevulinic Acid; Laser Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Arm 1 - ALA (Experimental): Patients receive topical ALA topical (aminolevulinic acid) 2 hours before PDT.
  Interventions: Drug: aminolevulinic acid
- Arm 2 (Experimental): Patients receive topical ALA topical (aminolevulinic acid) 4 hours before PDT
  Interventions: Drug: aminolevulinic acid
- Arm 3 (Experimental): Patients receive topical ALA (aminolevulinic acid) 24 hours before PDT. Each anatomic area is divided into subunits (e.g., right and left arm, right and left side of the face). The subunits are randomized to receive 1 or 2 pulses of the laser treatment
  Interventions: Drug: aminolevulinic acid
- Arm 4 (Experimental): Vbeam laser pulse (photodynamic therapy) is applied to the subunit
  Interventions: Procedure: laser therapy
- Arm 5 (Experimental): Vbeam laser pulses (photodynamic therapy) are applied to the subunit. Patients may receive up to 3 treatments (including pretreatment, ALA, and PDT) at least 1 month apart
  Interventions: Procedure: laser therapy

INTERVENTIONS:
Drug: aminolevulinic acid
  Arms: Arm 1 - ALA; Arm 2; Arm 3
Procedure: laser therapy
  Arms: Arm 4; Arm 5

SUMMARY:
RATIONALE: Photodynamic therapy uses a drug that becomes active when it is exposed to a certain kind of light. When the drug is active, abnormal cells are killed. Photodynamic therapy using topical aminolevulinic acid may be effective against actinic keratosis.

PURPOSE: This randomized clinical trial is studying how well different photodynamic therapy regimens using topical aminolevulinic acid work in treating patients with actinic keratosis.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine, using fluorescence measurements, the protoporphyrin IX (PpIX) accumulation in thin actinic keratoses (AK) and actinically damaged skin on the face, scalp, and upper torso (stratum 1) and the PpIX accumulation in thick AK and actinically damaged skin on the arms and legs (stratum 2) as a function of skin preparation, aminolevulinic acid (ALA) application time, and body site.
* To determine the extent that the PpIX is photobleached by the treatment light.

Secondary

* To assess the effects of different treatment conditions on acute reactions of AK and sun damaged skin to ALA-photodynamic therapy (PDT) occurring 24-48 hours after PDT.
* To assess the effects of different treatment conditions on the efficacy of ALA-PDT.
* To examine the histological response to ALA-PDT.
* To determine, using fluorescence measurements, the PpIX accumulation in incidental thick AK that may occur in stratum 1, and the PpIX accumulation in incidental thin AK that may occur in stratum 2 as a function of skin preparation, ALA application time and body site.
* To determine the extent that the PpIX in these incidental lesions is photobleached by treatment light.

OUTLINE: The randomization is a two-step restricted block process for application time and skin preparation, followed by randomization for light dose (1 vs 2 pulses) within the anatomic site. Within each stratum (stratum 1 or 2), lesions in each separate anatomic area (face and neck, scalp, upper torso; arms, legs) are randomized to receive 1 of 3 pretreatment skin preparation before receiving topical aminolevulinic acid (ALA): pretreatment with acetone, gentle abrading, or no pretreatment. Patients are randomized to receive ALA at different times before the photodynamic therapy (PDT).

* Arm I: Patients receive topical ALA 2 hours before PDT.
* Arm II: Patients receive topical ALA 4 hours before PDT.
* Arm III: Patients receive topical ALA 24 hours before PDT. Each anatomic area is divided into subunits (e.g., right and left arm, right and left side of the face). The subunits are randomized to receive 1 or 2 pulses of the laser treatment.
* Arm IV: 1 Vbeam laser pulse (photodynamic therapy) is applied to the subunit.
* Arm V: 2 Vbeam laser pulses (photodynamic therapy) are applied to the subunit. Patients may receive up to 3 treatments (including pretreatment, ALA, and PDT) at least 1 month apart. Patients with progressive lesions or lesions that have not responded after 3 treatments may receive diagnostic biopsy to check for invasive squamous cell carcinoma and referred to treatment off study.

Patients undergo biopsies at baseline, before and after ALA application prior to light treatment, and up to 24 hours after light treatment to analyze cytokines and genes specific to actinic keratoses.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Actinic keratosis lesion located in any of the following body sites:

  * Stratum 1*: face and neck, scalp, or upper torso

    * At least 1 clinically evident thin actinic keratosis on each side of the midline of any of the above areas
  * Stratum 2*: arms or legs

    * At least 1 clinically evident thick actinic keratosis on each arm or leg NOTE: *One patient may be in one or both strata depending on the location of the lesion(s)
* Lesions to be treated on this protocol must not have been previously treated by other modalities for at least 2 months prior to study entry

PATIENT CHARACTERISTICS:

* No porphyria or known hypersensitivity to porphyrins
* No known photosensitivity disease
* No known sensitivity to any components of aminolevulinic acid topical solution
* Not pregnant or nursing

PRIOR CONCURRENT THERAPY:

* Other concurrent topical therapies at lesion sites other than those used in this protocol are allowed
* No other concurrent photosensitizer drugs

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2005-05; Primary Completion 2009-01 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nathalie Zeitouni, MD,, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was activated prior to RPCI putting a centralize data entry and data management. Data entry of the treatment arm assignments and outcomes was done by PI's staff and has since been lost. The PI died and all attempts to retrieve the data have failed.
Groups:
- Unknown Trt Arm: Aminolevulinic Acid and Laser Therapy: Arm1: Patients receive topical ALA topical (aminolevulinic acid) 2 hours before PDT.
  Arm2: Patients receive topical ALA topical (aminolevulinic acid) 4 hours before PDT Arm 3: Patients receive topical ALA (aminolevulinic acid) 24 hours before PDT. Each anatomic area is divided into subunits (e.g., right and left arm, right and left side of the face). The subunits are randomized to receive 1 or 2 pulses of the laser treatment Arm 4: Vbeam laser pulse (photodynamic therapy) is applied to the subunit Arm 5: Vbeam laser pulses (photodynamic therapy) are applied to the subunit. Patients may receive up to 3 treatments (including pretreatment, ALA, and PDT) at least 1 month apart
Period: Overall Study
Arm/Group | Unknown Trt Arm: Aminolevulinic Acid and Laser Therapy
Started | 12
Completed | 7
Not Completed | 5
Not completed — Withdrawal by Subject | 5

BASELINE CHARACTERISTICS:
Population: All treated and eligible patients
Arm/Group | Unknown Trt Arm: Aminolevulinic Acid and Laser Therapy
Number analyzed (Participants) | 12
Age, Continuous [Median (Standard Deviation); unit: years] | 62.4 (15.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 6

OUTCOME MEASURES:

1. Primary Outcome: Protoporphyrin IX (PpIX) Accumulation as a Function of Skin Preparation, Aminolevulinic Acid Application Time, and Body Site
Population: Study was activated prior to RPCI putting a centralize data entry and data management. Data entry of the treatment arm assignments and outcomes was done by PI's staff and has since been lost. The PI died and all attempts to retrieve the data have failed.
Arm/Group | Unknown Trt Arm: Aminolevulinic Acid and Laser Therapy
Number analyzed (Participants) | 0

2. Primary Outcome: Extent That the PpIX is Photobleached by the Treatment Light
Population: as for outcome 1
Arm/Group | Unknown Trt Arm: Aminolevulinic Acid and Laser Therapy
Number analyzed (Participants) | 0

3. Secondary Outcome: Effects of Different Treatment Conditions on Acute Reactions of Actinic Keratoses (AK) and Sun Damaged Skin Occurring 24-48 Hours After Photodynamic Therapy
Population: as for outcome 1
Arm/Group | Unknown Trt Arm: Aminolevulinic Acid and Laser Therapy
Number analyzed (Participants) | 0

4. Secondary Outcome: Effects of Different Treatment Conditions on Efficacy
Population: as for outcome 1
Arm/Group | Unknown Trt Arm: Aminolevulinic Acid and Laser Therapy
Number analyzed (Participants) | 0

5. Secondary Outcome: Histological Response
Population: as for outcome 1
Arm/Group | Unknown Trt Arm: Aminolevulinic Acid and Laser Therapy
Number analyzed (Participants) | 0

6. Secondary Outcome: PpIX Accumulation in Incidental AK as a Function of Skin Preparation, Aminolevulinic Acid Application Time, and Body Site
Population: as for outcome 1
Arm/Group | Unknown Trt Arm: Aminolevulinic Acid and Laser Therapy
Number analyzed (Participants) | 0

7. Secondary Outcome: Extent That the PpIX is Photobleached by the Treatment Light in Incidental Lesions
Population: as for outcome 1
Arm/Group | Unknown Trt Arm: Aminolevulinic Acid and Laser Therapy
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Description: Study was activated prior to RPCI putting a centralize data entry and data management. Data entry was done by PI's staff. PI died and left incomplete data. Efficacy and safety data were not analyzed.
Arm/Group | Unknown Trt Arm: Aminolevulinic Acid and Laser Therapy
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
Study was activated prior to RPCI putting a centralize data entry and data management. Data entry of the treatment arm assignments and outcomes was done by PI's staff and has since been lost. PI died, all attempts to retrieve the data have failed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes